CLINICAL TRIAL: NCT01852825
Title: A Two Part, Randomized Clinical Trial to Study Biomarkers of MK-8237 (SCH 900237) Treatment in Subjects With House Dust Mite Induced Allergic Rhinitis or Rhinoconjunctivitis
Brief Title: MK-8237 (SCH900237) Biomarker Study in Participants With Allergic Rhinitis or Rhinoconjunctivitis (MK-8237-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 8237-009; 2012-005621-70 (EudraCT Number)
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NAC + MK-8237 (Part 2) (Experimental): Nasal Allergen Challenge (NAC) treatment consisting of 1800 Biological Units (BU) of HDM extract on Days -14, 56 and 84; starting on Day 1 a single tablet of MK-8237 with 12 Development Units (DUs), administered sublingually, at approximately the same time each day for 84 days (+/- 5 days)
  Interventions: Biological: MK-8237; Biological: NAC
- NAC + Placebo (Part 2) (Placebo Comparator): NAC treatment consisting of 1800 BU of HDM extract on Days -14, 56 and 84; starting on Day 1 a single placebo tablet administered sublingually, at approximately the same time each day for 84 days (+/- 5 days)
  Interventions: Other: Placebo; Biological: NAC
- NAC (Part 1) (Experimental): Nasal Allergen Challenge (NAC) consisting of 100 µl fixed volume of 10,000 biological units (BU) of HDM extract delivered with a Pfeiffer Bidose Nasal Delivery System (or equivalent) to each nostril for a total dose of 1800 BU at the start of Part 1
  Interventions: Biological: NAC

INTERVENTIONS:
Biological: MK-8237 — A single tablet of MK-8237 with 12 DU, administered sublingually, at approximately the same time each day for 84 days (+/- 5 days)
  Arms: NAC + MK-8237 (Part 2)
Other: Placebo — A single placebo tablet administered sublingually, at approximately the same time each day for 84 days (+/- 5 days)
  Arms: NAC + Placebo (Part 2)
Biological: NAC — 0.1 mL fixed volume of 10,000 BU/mL of HDM extract is delivered with a Pfeiffer Bidose Nasal Delivery System (or equivalent) to each nostril for a total dose of 1800 BU at the start of Part 1; and in Part 2 on Days -14, 56 and 84

SUMMARY:
The purpose of this study is to assess the effect on various biomarkers of treatment with MK-8237 in participants with allergic rhinitis or rhinoconjunctivitis. In Part 1 of the study healthy participants undergo nasal allergen challenge (NAC) with house dust mite (HDM) extract in order to verify the operational performance of NAC and associated sample collection methods. Part 2, the main study, is a placebo controlled, double blind study of participants with HDM-induced allergic rhinitis or rhinoconjunctivitis. The primary hypotheses are that the changes from baseline in post-allergen challenge HDM-specific Immunoglobulin G4 (IgG4) and Immunoglobulin E blocking factor (IgE-BF) are greater after treatment with MK-8237 than after treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* healthy participants
* has a Body Mass Index (BMI) =< 30 kg/m^2
* female of reproductive potential remains abstinent or uses two acceptable methods of birth control from 2 weeks before first allergen challenge to 2 weeks after last allergen challenge; alternatively hormonal contraception may be used.

Part 2:

* has a Body Mass Index (BMI) =< 38 kg/m^2
* has a clinical history of allergic rhinitis/rhinoconjunctivitis to HDM for at least one year, and used medication to relieve symptoms within the last year
* does not have asthma, or has mild controlled asthma not requiring regular use over the 12 months prior to screening of any corticosteroids
* female of reproductive potential remains abstinent or use two acceptable methods of birth control from 2 weeks before first allergen challenge to at least 2 weeks after last allergen challenge or last dose of study drug, whichever is longer
* has not smoked or used tobacco for the prior 6 months, and agrees not to during study

Exclusion Criteria:

Parts 1 and 2:

* is experiencing at the first NAC visit, symptoms from an upper or lower respiratory tract infection (viral or bacterial)
* has participated within the prior 3 months in another investigational study (that included an investigational drug or agent)
* is directly associated with the administration of the study or is related to the investigational study staff
* is mentally or legally incapacitated, has significant emotional problems or has a history of clinically significant psychiatric disorder within the past 5 years
* has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
* has a history of cancer
* has a history of significant intolerability to drugs or food
* is positive for hepatitis B surface antigen, hepatitis C antibodies or HIV
* had major surgery or lost 1 unit (500 mL) of blood within the prior 4 weeks
* has a clinical history of chronic sinusitis during the prior 2 years
* has any nasal condition (e.g. nasal polyposis) that could confound efficacy or safety assessments
* is pregnant or expects to conceive during the study period
* is a nursing mother
* consumes more than 3 glasses of alcoholic beverages per day
* regularly uses any illicit drug, or has a history of drug or alcohol abuse within the prior 6 months

Part 2 only:

* is experiencing allergic rhinoconjunctivitis exacerbation at Screening NAC
* consumes excessive daily amounts of caffeinated beverages
* has a known history of allergy, hypersensitivity or intolerance to investigational medicines
* is sensitized and regularly exposed to animal dander and molds in the home or workplace in a manner that might interfere with the study in the opinion of the investigator
* is sensitized and regularly exposed to seasonal allergens such as Birch or grass pollen (sensitized but out of season is acceptable however)
* has a history of chronic urticaria and/or angioedema within the prior 2 years
* has had previous immunotherapeutic treatment with any HDM allergen for more than 1 month during the prior 3 years
* is receiving any specific immunotherapy within prior 60 days
* has a history of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy due to an unknown cause or an inhalant allergen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2015-07-20 (Actual); Study Completion 2015-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gunawardana NC, Zhao Q, Carayannopoulos LN, Tsai K, Malkov VA, Selverian D, Clarke G, Mant T, Butts BD, Lund K, Hansel TT, Nolte H. The effects of house dust mite sublingual immunotherapy tablet on immunologic biomarkers and nasal allergen challenge symptoms. J Allergy Clin Immunol. 2018 Feb;141(2):785-788.e9. doi: 10.1016/j.jaci.2017.08.016. Epub 2017 Sep 11. No abstract available. PMID 28911971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1, healthy participants aged 18-55 years were enrolled; In Part 2, participants with house dust mite (HDM)-induced allergic rhinitis or rhinoconjunctivitis, aged 18-55, were enrolled.
Groups:
- NAC (Part 1): Nasal Allergen Challenge (NAC) treatment consisting of 100 µl fixed volume of 10,000 biological units (BU) of HDM extract delivered with a Pfeiffer Bidose Nasal Delivery System (or equivalent) to each nostril for a total dose of 1800 BU at the start of Part 1
Period: Overall Study
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Started | 16 | 7 | 3
Completed | 14 | 7 | 3
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1) | Total
Number analyzed (Participants) | 16 | 7 | 3 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (8.6) | 36.1 (13.2) | 25.7 (4.0) | 31.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 1 | 12
  Male | 8 | 4 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in D. Farinae HDM-specific IgG4 Antibodies in Serum at 12 Weeks (Part 2)
Description: Blood was collected from participants treated with Dermatophagoides (D.) farinae HDM and then with MK-8237 or placebo, and the amount of HDM-specific IgG4 antibodies in serum at baseline and at week 12 were measured. Fold change from baseline was evaluated based on constrained longitudinal data analysis (cLDA) method with log transformed data. The model included time (categorical variable), treatment, and time by treatment interaction as fixed effects and participants as random effect. Least squares geometric means are presented. It is hypothesized that the change from baseline is statistically greater with MK-8237 treatment than with placebo. This hypothesis is supported if the lower bound of the two-sided 90% confidence interval for the geometric mean fold difference is >1.0.
Time Frame: Baseline and 12 weeks
Population: All randomized participants from Part 2 who are compliant with the study procedures and have available data from at least one treatment. Participants from Part 1 were not analyzed because they were not treated with MK-8237 or placebo.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 14 | 7 | 0
Fold Change | 0.392 [0.249 to 0.615] | 0.166 [0.097 to 0.285] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); The hypothesis is supported if the lower bound of the two-sided 90% confidence interval for the Week 12 geometric mean fold difference is >1.0; Test type: Superiority or Other; p = 0.003, Constrained Longitudinal Data Analysis; Geometric Mean Ratio = 2.355, 90% CI 2-sided [1.515 to 3.661] — MK-8237 treatment divided by Placebo treatment

2. Primary Outcome: Change From Baseline in D. Pteronyssinus HDM-specific IgG4 Antibodies in Serum at 12 Weeks (Part 2)
Description: Blood was collected from participants treated with D. pteronyssinus HDM, and then with MK-8237 or placebo, and the amount of HDM-specific IgG4 antibodies in serum at baseline and at week 12 were measured. Fold change from baseline was evaluated based on cLDA method with log transformed data. The model included time (categorical variable), treatment, and time by treatment interaction as fixed effects and participants as random effect. Least squares geometric means are presented. It is hypothesized that the change from baseline is statistically greater with MK-8237 treatment than with placebo. This hypothesis is supported if the lower bound of the two-sided 90% confidence interval for the geometric mean fold difference is >1.0.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 14 | 7 | 0
Fold Change | 0.619 [0.397 to 0.966] | 0.284 [0.164 to 0.490] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, Constrained Longitudinal Data Analysis; Geometric Mean Ratio = 2.182, 90% CI 2-sided [1.364 to 3.490] — MK-8237 treatment divided by Placebo treatment

3. Primary Outcome: Change From Baseline in HDM-specific IgE Blocking Factor (IgE-BF) in Serum at 12 Weeks
Description: Blood was collected from participants treated with D. pteronyssinus and D.farinae HDM and then with either MK-8237 or placebo, and the amount of IgE-BF in serum was measured based on an Ordinary IgE measurement and an assay in the presence of Competitors; with IgE-BF = 1 - (Competitive IgE/Ordinary IgE). This ranges from 0 (no IgE blocked) to 1 (all IgE blocked); and as it is based on a ratio there are no units. Change from baseline (12 weeks minus baseline) was evaluated based on cLDA method, and was analyzed based on the original scale. The model included time (categorical variable), treatment, and time by treatment interaction as fixed effects and participants as random effect. It is hypothesized that the change from baseline is statistically greater with MK-8237 treatment than with placebo. This hypothesis is supported if the lower bound of the 1-tailed 95% CI around the 12 week mean difference in change from baseline in HDM-specific IgE blocking factor response excludes zero.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 14 | 7 | 0
Ratio | 0.097 [-0.032 to 0.226] | -0.141 [-0.317 to 0.035] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); The hypothesis is supported if the lower bound of the 1-tailed 95% CI around the mean difference in change from baseline excludes zero; Test type: Superiority or Other; p = 0.027, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = 0.238, 90% CI 2-sided [0.066 to 0.410] — MK-8237 treatment minus Placebo treatment

4. Secondary Outcome: Change From Baseline in 6.5 Hours Post-NAC Interleukin-5 (IL-5) Protein Concentration in Nasal Exudates Following 12 Weeks of Treatment (Part 2)
Description: Blood was collected from participants treated with D. pteronyssinus and D.farinae HDM and then with either MK-8237 or placebo, and the levels of Il-5 protein 6.5 hours after NAC in serum at baseline and at week 12 were measured. Fold change from baseline and between-treatment comparison was evaluated based on cLDA method with log transformed data. IL-5 protein concentration was measured in nasal exudates collected both pre- and post-nasal challenge. Least squares geometric means are presented.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Fold change
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 14 | 6 | 0
Fold change | 9.444 [3.852 to 23.153] | 8.843 [2.245 to 34.836] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); Test type: Superiority or Other; p = 0.935, Constrained Longitudinal Data Analysis; Geometric Mean Ratio = 1.068, 90% CI 2-sided [0.272 to 4.190] — MK-8237 treatment divided by Placebo treatment

5. Secondary Outcome: Change From Baseline in 6.5 Hours Post-NAC Nasal Epithelial Eosinophil-related Messenger RNA (mRNA) Signature Following 12 Weeks of Treatment (Part 2)
Description: Blood was collected from participants treated with D. pteronyssinus and D.farinae HDM and then with either MK-8237 or placebo, and the levels of nasal epithelial eosinophil-related mRNA signature 6.5 hours after NAC in serum at baseline and at week 12 were measured. The mRNA signature is derived from nine gene transcripts which were measured using the NanoString nCounter Gene Expression Assay. Positive control and pre-specified housekeeping gene normalization methods recommended by nSolver were used to normalize the transcripts. The average of the expression level of the nine genes was used to describe the eosinophil mRNA signature. Fold change from baseline and between-treatment comparison was evaluated based on cLDA method with log transformed data. Least squares geometric means are presented.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Fold change
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 9 | 4 | 0
Fold change | 2.618 [0.911 to 5.160] | 0.981 [0.267 to 3.610] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); Test type: Superiority or Other; p = 0.296, Constrained Longitudinal Data Analysis; Geometric Mean Ratio = 2.210, 90% CI 2-sided [0.605 to 8.066] — MK-8237 treatment divided by Placebo treatment

6. Secondary Outcome: Change From Baseline in Time Weighted Average (TWA) Over 1 Hour Pre-NAC Through 1 Hour Post-NAC Visual Analog Score (VAS) for Sneezing, Rhinorrhea, Congestion and Nasal Itch Following 12 Weeks of Treatment (Part 2)
Description: A visual analog scale (VAS) representing the spectrum of symptoms from absent (0) to extremely severe (100) for each of rhinorrhea, nasal blockage, sneezing and nasal itch were summed to obtain an overall score. The range of VAS overall score is 0 - 400, with higher numbers representing worse symptoms. The models for the time-weighted mean (TWA) of the summed scores over 1 hour pre-NAC through hour 1 following NAC were constructed at the original scale.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2) | NAC (Part 1)
Number analyzed (Participants) | 14 | 6 | 0
Score on a scale | 53.065 [25.797 to 80.334] | 114.180 [74.723 to 153.638] |
Statistical Analysis 1: Comparison: NAC + MK-8237 (Part 2) vs NAC + Placebo (Part 2); Test type: Superiority or Other; p = 0.014, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -61.115, 90% CI 2-sided [-100.185 to -22.045] — MK-8237 treatment minus Placebo treatment

ADVERSE EVENTS:
Time Frame: Part 1: Up to 17 days after treatment; Part 2: Up to 101 days after treatment
Description: All participants who received at least one dose of the investigational drug.
Arm/Group | NAC (Part 1) | NAC + MK-8237 (Part 2) | NAC + Placebo (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 0/3 | 14/16 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC (Part 1) (N=3) | NAC + MK-8237 (Part 2) (N=16) | NAC + Placebo (Part 2) (N=7)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 4 (8) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 3 (6) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Tongue pruritus (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 6 (7) | 4 (5)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.